CLINICAL TRIAL: NCT05947890
Title: A Phase 2a Clinical Trial to Evaluate the Safety and Immunogenicity of MTBVAC in Adolescents and Adults Living With and Without HIV in South Africa
Brief Title: Evaluating the Safety and Immunogenicity of MTBVAC in Adolescents and Adults Living With and Without HIV in South Africa
Acronym: HVTN605A5421
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Biofabri, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 605/A5421; UM1AI068614 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: HIV I Infection; Tuberculosis
Keywords: HIV; TB
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- 1.1a - Adolescents and adults without HIV and negative interferon-gamma release assay (Experimental): Participants will receive MTBVAC as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: MTBVAC
- 1.1b - Adolescents and adults without HIV and negative interferon-gamma release assay (Experimental): Participants will receive BCG as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: BCG
- 1.2a - Adolescents and adults without HIV and positive interferon-gamma release assay (Experimental): Participants will receive MTBVAC as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: MTBVAC
- 1.2b - Adolescents and adults without HIV and positive interferon-gamma release assay (Experimental): Participants will receive BCG as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: BCG
- 2.1 a- Adolescents and adults with well-controlled HIV and negative interferon-gamma release assay (Experimental): Participants will receive MTBVAC as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: MTBVAC
- 2.1.b - Adolescents and adults with well-controlled HIV and negative interferon-gamma release assay (Experimental): Participants will receive BCG as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: BCG
- 2.2 a- Adolescents and adults with well-controlled HIV and positive interferon-gamma release assay (Experimental): Participants will receive MTBVAC as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: MTBVAC
- 2.2 b- Adolescents and adults with well-controlled HIV and positive interferon-gamma release assay (Experimental): Participants will receive BCG as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: BCG
- 3.1 a- Adults with well-controlled HIV and negative interferon-gamma release assay (Experimental): Participants will receive MTBVAC as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: MTBVAC
- 3.1 b- Adults with well-controlled HIV and negative interferon-gamma release assay (Experimental): Participants will receive BCG as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: BCG
- 3.2 a- Adults with well-controlled HIV and positive interferon-gamma release assay (Experimental): Participants will receive MTBVAC as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: MTBVAC
- 3.2 b- Adults with well-controlled HIV and positive interferon-gamma release assay (Experimental): Participants will receive BCG as a 0.1 mL intradermal (ID) injection, in the upper arm once at Week 0.
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: MTBVAC — The MTBVAC vaccine is a freeze-dried lyophilized pellet containing live attenuated strain MTBVAC01 derived from Mycobacterium tuberculosis (M.tb). Excipients include sucrose and sodium glutamate.
  Arms: 1.1a - Adolescents and adults without HIV and negative interferon-gamma release assay; 1.2a - Adolescents and adults without HIV and positive interferon-gamma release assay; 2.1 a- Adolescents and adults with well-controlled HIV and negative interferon-gamma release assay; 2.2 a- Adolescents and adults with well-controlled HIV and positive interferon-gamma release assay; 3.1 a- Adults with well-controlled HIV and negative interferon-gamma release assay; 3.2 a- Adults with well-controlled HIV and positive interferon-gamma release assay
Biological: BCG — The active substance in BCG vaccine is a freeze-dried powder containing live attenuated Mycobacterium bovis BCG, Danish strain 1331 and sodium glutamate as a stabilizer. The powder is white and crystalline and may be difficult to see due to the small amount contained in each vial.
  Arms: 1.1b - Adolescents and adults without HIV and negative interferon-gamma release assay; 1.2b - Adolescents and adults without HIV and positive interferon-gamma release assay; 2.1.b - Adolescents and adults with well-controlled HIV and negative interferon-gamma release assay; 2.2 b- Adolescents and adults with well-controlled HIV and positive interferon-gamma release assay; 3.1 b- Adults with well-controlled HIV and negative interferon-gamma release assay; 3.2 b- Adults with well-controlled HIV and positive interferon-gamma release assay

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of MTBVAC in adolescents and adults living with and without HIV in South Africa

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of MTBVAC in adolescents and adults living with and without HIV in South Africa.

The study will be conducted in two parts (Part A and B). Part A will include two Cohorts (Cohort 1 and 2) and each Cohort will have four groups. Part B will have one Cohort which will also have four groups.

Participants will be recruited into three cohorts (Cohorts 1-3) based on their HIV status and, for People Living With HIV, their CD4+ T cell count and WHO clinical stage prior to ART initiation/re-initiation. Within each cohort, they will be stratified into subgroups based on their IGRA status.

For Cohorts 1 and 2 which will enroll simultaneously, participants will be randomized to receive MTBVAC or BCG according to the ratio of the planned sample sizes within the cohort; there is no placebo group in this trial.

Enrollment of Cohort 3 will proceed if safety criteria are met for Cohorts 1 and 2, with randomization to MTBVAC and BCG.

Participants in all groups will receive a single ID study product injection of 0.1 mL in volume and will be followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of 12 through 55 years, on the day of enrollment.
* Access to a participating HVTN or ACTG CRS and willingness to be followed for the planned duration of the study.
* For volunteers 18 years of age or older: ability and willingness to provide informed consent.
* For volunteers less than 18 years of age: parent or legal guardian is willing and able to provide informed consent for potential participant's study participation; in addition, when applicable per ethics committee policies and procedures, potential participant is willing and able to provide written assent for study participation.
* Assessment of Understanding (AoU): volunteer demonstrates understanding of this study and completes a questionnaire prior to vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly.
* Prior receipt of BCG vaccine in infancy as determined by the site investigator.
* Agrees not to enroll in another study of an investigational study product until after the last scheduled clinic visit. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 605/A5421 PSRT are required prior to enrollment into HVTN 605/A5421.
* Good general health as shown by medical history, physical exam, and screening laboratory tests and assessed by the site investigator.
* Willingness to receive HIV-related test results.
* For volunteers living without HIV:

  1. Negative HIV-1 and -2 blood test: Non-US sites may use locally available assays that have been approved by HVTN Laboratory Operations
  2. Assessed by the clinic staff as having a low likelihood of acquiring HIV and is committed to maintaining behavior that is consistent with a lower likelihood of acquiring HIV through the last required protocol clinic visit
  3. Willingness to discuss their potential for HIV acquisition and is amenable to HIV risk reduction counseling
* For volunteers living with HIV:

  1. For both Cohorts 2 and 3: Completed one course of tuberculosis preventive treatment (TPT) as determined by the site investigator.

     Documented HIV viral suppression (Plasma HIV levels < 50 copies/mL) collected at least three months and up to 15 months prior to enrollment (with no intervening HIV-1 RNA results ≥ 50 copies/mL) and from screening labs.

     Has been receiving at least 6 months of ART prior to enrollment, as determined by the site investigator
  2. For Cohort 2: WHO HIV clinical stage 1 or 2 prior to initiation (or re-initiation in case of treatment interruption/default) of ART.

CD4+ T-cell count of ≥ 200 cells/mm3 (during screening) 3. For Cohort 3: Advanced HIV disease (defined as CD4 count less than 200 cells/mm3 or WHO HIV clinical stage 3 or 4) prior to initiation (or re-initiation) of ART. Advanced HIV defined as CD4 count less than 200 cells/mm3 or WHO stage 3 or 4. Current CD4+ T-cell count of ≥ 100 cells/ mm3 (during screening)

* Laboratory Inclusion Values - Has normal or Grade 1 results of all of the following at screening:

Hemoglobin (≥ 9.5 g/dL or ≥ 5.88 mmol/L for males and females less than 13 years of age; ≥ 9.5 g/dL or ≥ 5.88 mmol/L for females 13 years of age and older; ≥ 10.0 g/dL or ≥ 6.19 mmol/L for males 13 years of age and older); White blood cell count (≥ 2000 cells/mm3 or ≥ 2.000 × 109 cells/L); Platelet count (≥ 100,000 cells/mm3 or ≥ 100.000 × 109 cells/L); Creatinine (≤ 1.3 × upper limit of normal [ULN]); Alanine aminotransferase (ALT) (< 2.5 × ULN); Aspartate aminotransferase (AST) (< 2.5 × ULN)

* Negative Hepatitis B surface antigen (HBsAg).
* Negative anti-Hepatitis C virus Abs (anti-HCV), or negative HCV nucleic acid test if the anti-HCV is positive
* For volunteers assigned female sex at birth (AFAB) or intersex at birth and are of reproductive potential (hereafter referred to as "of pregnancy potential"): negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test at screening (ie, prior to randomization) and prior to study product administration on the day of study product administration. Persons who are NOT of pregnancy potential including having reached menopause (no menses for 1 year) or having undergone hysterectomy or bilateral oophorectomy, or tubal ligation (verified by medical records) are not required to undergo pregnancy testing.
* Reproductive status: A volunteer of pregnancy potential:

  1. Must agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until 10 weeks after vaccination.
  2. Volunteers of pregnancy potential must also agree not to seek pregnancy through alternative methods, such as artificial insemination, or in vitro fertilization until 10 weeks after vaccination.
  3. Volunteers of pregnancy potential must also agree not to undergo oocyte retrieval.

Exclusion Criteria:

* Weight less than 40 kg
* Known significant exposure to TB or receipt of tuberculin skin test in the six months prior enrollment, as determined by the site investigator based on potential participant/parent/guardian report and available medical records. [Note: Significant exposure is defined as close contact with a person who has active TB and has not completed TB treatment. Close contact is defined as sleeping in the same contiguous house/dwelling, and/or working or socializing in close proximity in an enclosed space frequently (eg, several times a week).]
* History of prior active TB disease, as determined by the site investigator based on participant/parent/guardian report and available medical, laboratory or radiographic records.
* Evidence of active TB disease as determined by the site investigator based on participant/parent/guardian report and available medical records, results from physical examination, two-view chest X-ray, and M.tb nucleic acid testing from an expectorated sputum, including a review of any available radiography; and, for volunteers living with HIV and a CD4 count <200 cells/mm3, a positive urine LAM test.
* Receipt of TB preventive therapy within 28 days prior to enrollment or expected to initiate TB preventive therapy during the study as determined by the site investigator based on participant/parent/guardian report and available medical records Note: Clinical indication for receipt of TB preventive therapy will be determined by the site investigator consistent with local standard guidelines. Potential participants on TB preventive therapy during screening may be enrolled once the exclusionary timeframes indicated above have elapsed. If the screening period is exceeded while this requirement is being met, a new screening attempt should be initiated.
* For volunteers living with HIV: current active AIDS-defining condition as determined by the site investigator based on participant/parent/guardian report and available medical records
* Blood products received within 120 days before vaccination.
* Investigational study products (non-vaccine) received within 28 days before vaccination.
* Pregnant or breastfeeding.
* Investigational TB vaccine(s) received in a prior TB vaccine trial or BCG vaccination outside infancy. For volunteers who have received control/placebo in a TB vaccine trial, the HVTN 605/A5421 PSRT will determine eligibility on a case-by-case basis.
* Investigational non-TB vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 605/A5421 PSRT for vaccines that have subsequently undergone licensure by the FDA or by the national regulatory authority where the volunteer is enrolling. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 605/A5421 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 1 years ago, eligibility for enrollment will be determined by the HVTN 605/A5421 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 28 days before first vaccination or scheduled within 28 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine).
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B).
* Allergy treatment with antigen injections within 28 days before first vaccination or that are scheduled within 14 days after first vaccination.
* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment).
* Serious adverse reactions to vaccines or to vaccine components including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a non-anaphylactic adverse reaction to pertussis vaccine as a child).
* Immunoglobulin received within 90 days before vaccination.
* Autoimmune disease, current or history (Not exclusionary: mild, well-controlled psoriasis)
* Immunodeficiency (Not exclusionary: HIV).
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  1. A process that would affect the immune response,
  2. A process that would require medication that affects the immune response,
  3. Any contraindication to repeated injections or blood draws,
  4. A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  5. A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  6. Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent, including but not limited to clinically significant substance or alcohol use disorder.
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Asthma exclusion criteria:

Asthma is exclusionary if the participant has ANY of the following:

1. Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR 2. Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR 3. Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR 4. Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.

* Diabetes mellitus type 1 or type 2. (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes. For these cases, control should be confirmed with an appropriate laboratory test (eg, fasting glucose, HbA1c) based on a specimen collected during screening.)
* Hypertension:

  1. If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently < 140 mm Hg systolic and < 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be < 140 mm Hg systolic and < 90 mm Hg diastolic at enrollment.
  2. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
* Bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study).
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen.
* History of angioedema or anaphylaxis (Not exclusionary: angioedema or anaphylaxis with known trigger and no episodes within five years.)
* History of generalized urticaria within past five years.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of unsolicited adverse events | Through study week 48
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Number of solicited adverse events | Through study week 16
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Number of Grade 3 or higher adverse events | Through study week 48
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Number of serious adverse events | Through study week 48
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Frequency and response of MTBVAC-reactive CD4+ cells expressing Th1 and/or Th17 cytokines | At baseline and study weeks 4
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of MTBVAC-reactive CD4+ cells expressing Th1 and/or Th17 cytokines | At baseline and study weeks10
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of MTBVAC-reactive CD8+ T cells expressing Th1 and/or Th17 cytokines | At baseline and study weeks 4
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of MTBVAC-reactive CD8+ T cells expressing Th1 and/or Th17 cytokines | At baseline and study weeks10
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells

SECONDARY OUTCOMES:
Number of unsolicited adverse events | Through study week 48
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Number of solicited adverse events | Through study week 16
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Number of Grade 3 or higher adverse events | Through study week 48
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Number of serious adverse events | Through study week 48
  Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
Frequency and response of BCG-reactive CD8+ T cells expressing Th1 and/or Th17 cytokines | At baseline and study week 4
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of BCG-reactive CD8+ T cells expressing Th1 and/or Th17 cytokines | At baseline and study week 10
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of BCG-reactive CD4+ expressing Th1 and/or Th17 cytokines | At baseline and study week 10
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of BCG-reactive CD4+ T cells expressing Th1 and/or Th17 cytokines | At baseline and study week 10
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of MTBVAC-reactive and BCG reactive CD8+ T cells expressing Th1 and/or Th17 cytokines | At study weeks 24 and 48
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
Frequency and response of MTBVAC-reactive and BCG reactive CD4+ T cells expressing Th1 and/or Th17 cytokines | At study weeks 24 and 48
  Measured by intracellular cytokine staining (ICS) and flow cytometry on cryopreserved peripheral blood mononuclear cells
MTBVAC-reactive and BCG-reactive IgA, IgG, and IgM binding Abs | At baseline and study weeks 4, 10, 24, and 48
  Measured using binding antibody multiplex assay (BAMA)
Gene expression profiles to evaluate innate immunogenicity in response to MTBVAC vaccination | At baseline and study weeks 1, 4, and 10
  Measured by RNA-seq in whole blood
Gene expression profiles to evaluate innate immunogenicity in response to BCG revaccination | At baseline and study weeks 1, 4, and 10
  Measured by RNA-seq in whole blood
Whole blood phenotyping to evaluate innate immunogenicity in response to MTBVAC vaccination | At baseline and study weeks 1, 4, and 10
  Measured by flow cytometry
Whole blood phenotyping to evaluate innate immunogenicity in response to BCG revaccination | At baseline and study weeks 1, 4, and 10
  Measured by flow cytometry
Measurement of soluble proinflammatory mediators in serum to evaluate innate immunogenicity in response to MTBVAC vaccination | At baseline and study weeks 1, 4, and 10
  Measure by multiplex protein detection assays and/or enzyme-linked immunosorbent assay (ELISA)
Measurement of soluble proinflammatory mediators in serum to evaluate innate immunogenicity in response to BCG revaccination | At baseline and study weeks 1, 4, and 10
  Measure by multiplex protein detection assays and/or enzyme-linked immunosorbent assay (ELISA)
Acceptability of the study products to assess the acceptability of MTBVAC vaccination | At study week 24 and the last scheduled clinic visit
  Scores derived from questionnaire responses Derived from questionnaire responses
Acceptability of the study products to assess the acceptability of BCG revaccination | At study week 24 and the last scheduled clinic visit
  Scores derived from questionnaire responses Derived from questionnaire responses

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, Study Chair — South African Tuberculosis Vaccine Initiative; Limakatso Lebina, Study Chair — Africa Health Research Institute (AHRI)
Locations (16):
- South Africa (16):
  - Soweto - Gauteng, Johannesburg, Gauteng
  - Johannesburg - CHRU, Westdene, Gauteng
  - Durban - Botha's Hill CRS, Durban, KwaZulu-Natal
  - Durban - Wentworth, Durban, KwaZulu-Natal
  - Cape Town - UCTLI, Cape Town, Western Cape
  - Cape Town - Emavundleni, Cape Town, Western Cape
  - Cape Town - Groote Schuur, Cape Town, Western Cape
  - Worcester - SATVI, Worcester, Western Cape
  - Cape Town - Khayelitsha, Cape Town
  - Durban - Chatsworth, Chatsworth
  - Durban eThekwini, Durban
  - Durban - Isipingo, Isipingo
  - Klerksdorp, Klerksdorp
  - Ladysmith, Ladysmith
  - Rustenburg CRS, Rustenburg
  - Soshanguve, Soshanguve